CLINICAL TRIAL: NCT02826590
Title: The Effects of Spinal Mobilizations on Symptoms, Neck 3D Movement, Neck Muscle Electromyography and Sympathetic Nervous System Activity in People With Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016/066
Record Dates: First submitted 2016-06-14; First posted 2016-07-11 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neck passive mobilizations (Experimental): Neck passive mobilizations
  Interventions: Other: Neck passive mobilizations
- Manual contact (Placebo Comparator): Manual contact
  Interventions: Other: Manual contact

INTERVENTIONS:
Other: Neck passive mobilizations — Passive mobilizations performed to the neck of the participant by a Physiotherapist
  Arms: Neck passive mobilizations
Other: Manual contact — Manual contact applied to the neck of the participant by a Physiotherapist
  Arms: Manual contact

SUMMARY:
This study investigates the effects of spinal mobilizations on symptoms, 3D movement of the neck, neck muscle electromyography and sympathetic nervous system activity in people with neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Intermittent neck pain
* That worsens or improves with certain neck movements or positions
* Has not been caused by a blow, fall or accident

Exclusion Criteria:

* Cervicobrachialgia
* Has been treated with or is awaiting neck surgery
* Diagnosed with a particular inflammatory disease or spinal condition
* Where treatment with cervical mobilizations is contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-06; Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Change in muscle activity assessed by neck muscle electromyography | Baseline and 2 minutes after intervention
Change in 3D neck movement assessed with a 10 camera Vicon system | Baseline and 2 minutes after intervention
Change in sympathetic nervous system activity assessed by measuring right hand finger temperature | Baseline for 2 minutes immediately before intervention, during intervention (15 minutes) and for 2 minutes immediately after intervention
  Measurement unit: degrees celsius
Change in sympathetic nervous system activity assessed by measuring right hand finger galvanic response | Baseline for 2 minutes immediately before intervention, during intervention (15 minutes) and for 2 minutes immediately after intervention
  Measurement unit: microsiemens
Global rating of change scale | Baseline and 10 minutes after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Atlas Fisioterapia, Donostia / San Sebastian, Gipuzkoa, Spain

IPD SHARING:
Plan to Share IPD: Undecided